CLINICAL TRIAL: NCT04195607
Title: Epidemiological Profile of Children With Early Caries: a Study in the Hauts-de-France Region
Brief Title: Epidemiological Profile of Children With Early Caries.
Acronym: EPIECC
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RNI_2018_97; 2019-A00827-50 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to determine the different profiles of patients with early caries consulting at the Lille CHU and to analyse the characteristics associated with the severity of the pathology. The data will be collected using a simple clinical examination of the child and a survey of the parent using a questionnaire. The typology of patients with early caries will be analysed according to the predefined variables collected using the questionnaire via a main component analysis in order to study the links between these variables. At the same time, a hierarchical classification analysis will be carried out to study the existence of homogeneous sub-groups of individuals in regard to the early caries. These sub-groups will be described

ELIGIBILITY:
Inclusion Criteria:

* be a child under the age of 6,
* having been diagnosed with early caries
* be accompanied by at least one parent (the mother or father).
* be affiliated to a social security

Exclusion Criteria:

* be a child over the age of 6

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with early caries who consult at the CHU in Lille.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of the image that parents have of dental health and carious disease | at day one
  Socio-demographic characteristics : country of birth of child, age of mother, country of birth of mother, level of education of mother (INSEE classification), occupation of mother (INSEE classification), maternal employment status (INSEE classification) , father's age, father's country of birth, father's educational level (INSEE classification), father's occupation (INSEE classification), father's work status (INSEE classification), number of children, number of people in same home, sibling rank with cavities, , distance between home and hospital.
Evaluation of the image that parents have of dental health and carious disease | at day one
  Parents' dental health knowledge : success score on a series of 7 questions about Oral Health Knowledge.
Evaluation of the image that parents have of dental health and carious disease | at day one
  Parental self-efficacy in dental health : evaluating the feeling of self-efficacy using a pass score on a series of 10 oral health questions.
Evaluation of the image that parents have of dental health and carious disease | at day one
  dental health behaviours of parents : success score on a series of 7 questions about oral health knowledge.
Evaluation of the image that parents have of dental health and carious disease | at day one
  Insurance, use, cost of care and modalities/use of pediatric dental care : social assistance, history of dental consultations in cities, number of practitioners consulted, difficulties in finding appropriate dental care for children, reason for consultation, renunciation of dental care for parent or child and reason, type of health coverage, cost of care.
Evaluation of the image that parents have of dental health and carious disease | at day one
  Locus of control in parental dental health : assessment using a simple question: "do you think you are personally responsible for the presence of caries in your child".
Evaluation of the image that parents have of dental health and carious disease | at day one
  Perceived importance of dental health behaviours among parents : evaluating the perceived importance of health behaviors using a score on a series of 14 oral health questions.
Evaluation of the image that parents have of dental health and carious disease | at day one
  Parents' dental health beliefs : evaluating the parents' dental health beliefs using a score on a series of 17 oral health questions.
Evaluation of the image that parents have of dental health and carious disease | at day one
  Distress of parents : evaluation using a series of 6 questions
Evaluation of the image that parents have of dental health and carious disease | at day one
  Chronic stress of parents : evaluation using a series of 2 questions.
Evaluation of the image that parents have of dental health and carious disease | at day one
  Social support : "how many people around you can count on when needed".
Evaluation of the image that parents have of dental health and carious disease | at day one
  Discrimination perceived by parents : evaluation using a response score to the 7 questions asked.
Evaluation of the image that parents have of dental health and carious disease | at day one
  Health literacy : evaluated using a single-question answer.
Evaluation of the image that parents have of dental health and carious disease | at day one
  Alcohol use among parents : evaluated using a three-question answer on frequency of alcohol consumption and quantity.

SECONDARY OUTCOMES:
frequency of patients with severe early caries in patients with early caries. | at day one
  Number of children with early stage severe caries according to the criteria of the American Academy of Pediatric Dentistry
Caries severity will be defined by the Severe Early Childhood Caries (S-ECC) | at day one
  This term is used if at least one of the following conditions is met:
  * Smooth surfaces of teeth are affected in a child under 3 years of age;
  * There is one or more caried anterior tooth(s), missing due to caries or fillings
  * The caod index* > 4 to 3 years, > 5 to 4 years or >6 to 5 years: the caod index indicates the number of temporary teeth decayed, absent due to caring or filling. It is between 0 and 20

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marquillier, DDS, Principal Investigator — University Hospital, Lille
Locations (1):
- Service d'Odontologie CHU, Lille, France

REFERENCES:
- [Result] Craquelin M, Trentesaux T, Delfosse C, Duhamel C, Matteucci R, Nonclercq S, Duhr A, Leblanc A, Behal H, Tiertant E, Lombrail P, Azogui-Levy S, Marquillier T. Family profiles in relation to early childhood caries: a cross-sectional study in France. BMJ Open. 2025 Jun 26;15(6):e100286. doi: 10.1136/bmjopen-2025-100286. PMID 40578875